CLINICAL TRIAL: NCT06768047
Title: Microporous Tape and Post Surgical Scars
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hagar Mohammed Hashem Elgarahy, Physical therapist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Microporous tape and scars
Record Dates: First submitted 2024-12-23; First posted 2025-01-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Microporous Tape; Hypertrophic Scars
Keywords: Microporous tape; Post surgical hypertrophic scars; Modified Vancouver Scar Scale; Schiotz tonometer.
MeSH Terms: conditions — Cicatrix, Hypertrophic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study group: receive Microporous tape and traditional physical therapy treatment (Active Comparator)
  Interventions: Other: Microporous tape; Other: Tradition physical therapy
- Control group receive traditional therapy ( (deep friction massage and stretching exercises) (Other)
  Interventions: Other: Tradition physical therapy

INTERVENTIONS:
Other: Microporous tape — Microporous tape is a dressing tape that was discovered to have scar modulating effects. It is made up of a conformable, inextensible, nonwoven fabric manufactured from 100% viscose and coated with a layer of acrylic adhesive. It is cheap, cost-effective, readily available, and relatively affordable for post surgical patients.
  Arms: Study group: receive Microporous tape and traditional physical therapy treatment
Other: Tradition physical therapy — Tradition physical therapy as stretching exercises and deep friction massage, Stretching is a form of physical exercise in which a specific muscle or tendon (or muscle group) is deliberately expanded and flexed in order to improve the muscle's felt elasticity and achieve comfortable muscle tone. The result is a feeling of increased muscle control, flexibility, and range of motion.
  Deep friction massage also known as cross friction massage, is a specific connective tissue massage which maintain the mobility within the soft tissue structures of ligament, tendon, and muscle, and prevent adherent scars from forming.

SUMMARY:
The aim of this study is to determine the effect of microporous taping on improving scar characteristics in post-surgical HTS.

DETAILED DESCRIPTION:
A scar can be defined as a mark or a blemish resulting from a healed wound. Scars are an integral part of human existence. All surgical incisions give rise to scars. Some scars are thin lines which are almost unnoticeable, whereas others become hypertrophic scars or keloids. Mechanical forces including tension have been shown to influence scarring as demonstrated in animal models and clinical experience. Wounds closed with excess tension are known to produce more scar tissue.A normal scar is characterized by minimal fibrosis; it is thin, flat and has a good colour match with the surrounding skin without distortion of the adjacent tissue. A scar is however considered abnormal when the amount of fibrosis is excessive or suboptimal or when it causes functional disability, psychosocial trauma or aesthetic distress to the patient. The conversion of normal scarring to hypertrophic scarring or the apparent overgrowth of scar support especially with the use of tape is critical during this period when increased tension across the scar would result in exaggerated scarring. The good management of scars is very important for patient to solve these consequences. Hypertrophic scars have seven times greater collagen production than normal due to increasing in collagenase activity. The hypertrophic scar develops at the third stage of wound healing. Scar maturation or remodeling lasts from three weeks to six months but may last for years.

The hypertrophic scars usually lead to connective tissue and muscles contracture resulting in limited R.O.M at the area of the scar Hypertrophic scars and keloids are Overgrowth of fibrous tissue that usually develop after healing of a skin injury and extend beyond the 2 original defect.

They often occur after local skin trauma as lacerations and burn injuries. Scarring following surgery or trauma is difficult to predict and physicians are highly concerned with minimizing scar appearance and value even small improvements in scarring as clinically meaningful.

to hypertrophic scarring or the apparent overgrowth of scar support especially with the use of tape is critical during this period when increased tension across the scar would result in exaggerated scarring. Hypertrophic scars cause cosmetic, psychological, physical (pain, and disabilities),financial and social consequences in addition to that , Hypertrophic scars lead to hypo-mobility ,connective tissue and muscles contracture.

The good management of scars is very important for patient to solve these consequences

.Hypertrophic scars have seven times greater collagen production than normal due to increasing in collagenase activity. The hypertrophic scar develops at the third stage of wound healing. Scar maturation or remodeling lasts from three weeks to six months but may last for years . The hypertrophic scar usually lead to connective tissue and muscles contracture resulting in limited R.O.M at the area of the scar Hypertrophic scars and keloids are Overgrowth of fibrous tissue that usually develop after healing of a skin injury and extend beyond the 2 original defect. They often occur after local skin trauma as lacerations and burn injuries . Scarring following surgery or trauma is difficult to predict and physicians are highly concerned with minimizing scar appearance and value even small improvements in scarring as clinically meaningful.

ELIGIBILITY:
Inclusion Criteria:

1. The patients' age will range from 20-45 years, and will be selected from both genders .
2. All patients will have hypertrophic scars after surgeries.
3. The general size of the scars will range from 5 to 7 cm'2

Exclusion Criteria:

1. The patients who will excluded from the study including those with infected post-operative wounds .
2. The patients whose wounds were closed secondarily or healed by secondary intention.
3. patients who are keloid formers.
4. Uncontrolled diabetes mellitus
5. Uncontrolled hypertension.
6. The patients who had a deep venous thrombosis (DVT).
7. Hypersensitivity reaction to Microporous tape.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-01-07 (Estimated); Primary Completion 2025-03-07 (Estimated); Study Completion 2025-03-07 (Estimated)

PRIMARY OUTCOMES:
Scars pliability | 8 weeks
  A Schiotz tonometer device (Riester, Germany, 0124) is simple to use, in expensive, reliable, requires little time to maintain and does not require supply of batteries or electricity. It has a free-floating, rod-like plunger with a 5.5 gm weight attached fits inside the barrel and other weights (7.5 or 10 grams) are put that can be equipped to the plunger. A Schiotz tonometer device was used as an objective device to assess the hypertrophic scar's pliability and elasticity

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Agrawal A, Ding J, Agrawal B, Kwan PO, Tredget EE. Stimulation of toll-like receptor pathways by burn eschar tissue as a possible mechanism for hypertrophic scarring. Wound Repair Regen. 2021 Sep;29(5):810-819. doi: 10.1111/wrr.12940. Epub 2021 May 27. PMID 34043867
- [Background] Ogawa R, Akaishi S, Huang C, Dohi T, Aoki M, Omori Y, Koike S, Kobe K, Akimoto M, Hyakusoku H. Clinical applications of basic research that shows reducing skin tension could prevent and treat abnormal scarring: the importance of fascial/subcutaneous tensile reduction sutures and flap surgery for keloid and hypertrophic scar reconstruction. J Nippon Med Sch. 2011;78(2):68-76. doi: 10.1272/jnms.78.68. PMID 21551963
- See also: Related Info — https://doi.org/10.21608/mjcu.2018.57135